CLINICAL TRIAL: NCT05425238
Title: Effects of Blood Flow Restriction Resistance Exercise on Strength and Transfer in Lower Cervical Spinal Cord Injury Patients
Brief Title: Blood Flow Restriction Resistance Exercise in Lower Cervical Spinal Cord Injury Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/22/0222
Record Dates: First submitted 2022-06-15; First posted 2022-06-21 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Cervical Spinal Cord Injury
MeSH Terms: interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blood flow restriction (Experimental): Resistance training protocol but with Blood flow restriction technique Standard BFR Application: a standard pressure (used for all patients) for e.g. 180 mmHg; a pressure relative to the patient's systolic blood pressure, for e.g. 1.2 - or 1.5-fold greater than systolic blood pressure.
  Interventions: Other: Blood flow restriction
- Conventional physical therapy (Active Comparator): Resistance training to stimulate skeletal muscle hypertrophy and strength adaptations in Duration of 6 weeks
  Interventions: Other: Conventional physical therapy

INTERVENTIONS:
Other: Blood flow restriction — strengthening protocol but with Blood flow restriction technique
  .Standard BFR Application: a standard pressure (used for all patients) for e.g. 180
  mmHg; a pressure relative to the patient's systolic blood pressure, for e.g. 1.2 - or 1.5-fold greater than systolic blood pressure.40% cuff pressure as percentage of LOP.(4) And performing BFR-RE with low load exercises. So 30% of 1 RPM would be enough 4 times a week for 6 week
  Arms: Blood flow restriction
Other: Conventional physical therapy — Resistance exercise 75 repetitions across four sets of exercises, with30 repetitions in the first set and 15 repetitions in each subsequent set. 4 times a week for 6
  Arms: Conventional physical therapy

SUMMARY:
This study is conducted to investigate the effects of low load Blood Flow Resistance exercise to improve strength and transfer in lower cervical spinal cord injury patientsCervical Spinal Cord injury patients have very less window of opportunity towards functional mode of life. In complete cervical spinal cord injuries only few muscles of upper limb are completely innervated and it is a need to gain maximum output and advantage out of that. Through conventional strength training it is possible to make him do unsupported sitting and transfer But with BFR-RE it may have a possibility to do this procedure in less time than the conventional strength training and patient will save cost of hospital stay as he may timely discharge from hospital early

ELIGIBILITY:
Inclusion Criteria:

* Both male and female, with age between 16-50 years.
* Patients evaluated with C6 to C8 tetraplegic complete injury.
* Patients classified in ASIA A, ASIA B.
* At least Muscle grading of grade 2.
* Patients with sub-acute, chronic stage.

Exclusion Criteria:

* Patients with other neurologic conditions, orthopedic problems, and uncontrolled metabolic diseases.
* Patients with muscles strength grading of less than 2.
* Undergone nerve transfer surgery.
* Patients with acute stage.
* History of DVT.
* Patients who are already performing structured physical activities such as muscle Strengthening exercises.

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2022-05-15 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
VAS- Visual Analogue Scale | 6th week
  To measure the intensity of pain
MAS- Modified Ashworth Scale | 6th week
  To measure the muscular hypertrophy and increased tone. Usually used to measure increased tone in spasticity but also used to measure hypertrophy resulted from normal muscles adaptations.
QIF-SF -- Quadriplegia Index Of Functionality-Small Form | 6th week
  To the transfer and functional ability in tetraplegic patients.
Hand Held Dynamometer | 6th week
  To measure the strength objectively and To measure the minor but notable changes in strength change which cannot be detected by MMT

CONTACTS AND LOCATIONS:
Overall Officials: Binash Afzal, PHD*, Principal Investigator — Riphah international university lahore campus
Locations (1):
- Lahore general Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roberts TT, Leonard GR, Cepela DJ. Classifications In Brief: American Spinal Injury Association (ASIA) Impairment Scale. Clin Orthop Relat Res. 2017 May;475(5):1499-1504. doi: 10.1007/s11999-016-5133-4. Epub 2016 Nov 4. No abstract available. PMID 27815685
- [Background] Kozlowski AJ, Heinemann AW. Using individual growth curve models to predict recovery and activities of daily living after spinal cord injury: an SCIRehab project study. Arch Phys Med Rehabil. 2013 Apr;94(4 Suppl):S154-64.e1-4. doi: 10.1016/j.apmr.2012.11.050. PMID 23527771
- [Background] Loenneke JP, Wilson JM, Marin PJ, Zourdos MC, Bemben MG. Low intensity blood flow restriction training: a meta-analysis. Eur J Appl Physiol. 2012 May;112(5):1849-59. doi: 10.1007/s00421-011-2167-x. Epub 2011 Sep 16. PMID 21922259
- [Background] Hughes L, Paton B, Rosenblatt B, Gissane C, Patterson SD. Blood flow restriction training in clinical musculoskeletal rehabilitation: a systematic review and meta-analysis. Br J Sports Med. 2017 Jul;51(13):1003-1011. doi: 10.1136/bjsports-2016-097071. Epub 2017 Mar 4. PMID 28259850
- [Background] Yasuda T, Fukumura K, Iida H, Nakajima T. Effect of low-load resistance exercise with and without blood flow restriction to volitional fatigue on muscle swelling. Eur J Appl Physiol. 2015 May;115(5):919-26. doi: 10.1007/s00421-014-3073-9. Epub 2014 Dec 10. PMID 25491331
- [Background] Anderson K, Aito S, Atkins M, Biering-Sorensen F, Charlifue S, Curt A, Ditunno J, Glass C, Marino R, Marshall R, Mulcahey MJ, Post M, Savic G, Scivoletto G, Catz A; Functional Recovery Outcome Measures Work Group. Functional recovery measures for spinal cord injury: an evidence-based review for clinical practice and research. J Spinal Cord Med. 2008;31(2):133-44. doi: 10.1080/10790268.2008.11760704. PMID 18581660
- [Background] Perwaiz S, Afzal MW, Fatima G. Comparison between qualitative and quantitative measurement of strength deficit in shoulder flexors of young females: A cross- sectional study. J Pak Med Assoc. 2021 Nov;71(11):2559-2562. doi: 10.47391/JPMA.011431. PMID 34783737
- [Background] Patterson SD, Hughes L, Warmington S, Burr J, Scott BR, Owens J, Abe T, Nielsen JL, Libardi CA, Laurentino G, Neto GR, Brandner C, Martin-Hernandez J, Loenneke J. Blood Flow Restriction Exercise: Considerations of Methodology, Application, and Safety. Front Physiol. 2019 May 15;10:533. doi: 10.3389/fphys.2019.00533. eCollection 2019. PMID 31156448
- [Background] Tuncali B, Karci A, Tuncali BE, Mavioglu O, Ozkan M, Bacakoglu AK, Baydur H, Ekin A, Elar Z. A new method for estimating arterial occlusion pressure in optimizing pneumatic tourniquet inflation pressure. Anesth Analg. 2006 Jun;102(6):1752-7. doi: 10.1213/01.ane.0000209018.00998.24. PMID 16717321